CLINICAL TRIAL: NCT01348334
Title: Use Of Three Types Of Synthetic Mesh Materials In Sling Surgery: A Prospective Randomized Clinical Trial Evaluating Effectiveness And Complications
Brief Title: Synthetic Mesh Materials In Sling Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Emrah Okulu, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ataturk TRH-01
Record Dates: First submitted 2011-04-28; First posted 2011-05-05 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2004-07

CONDITIONS: Incontinence
Keywords: Sling surgery; synthetic meshes; ultrapromesh®; mix mesh; incontinence; The Ultrapromesh® synthetic sling procedures have lower complications incidence and higher success rates than the other synthetic slings in 3-year follow-up.

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vypromesh®(Ethicon,USA) (Active Comparator): Vypromesh®(semiabsorbable multiflament mesh;non-absorbable Polypropylene+absorbable Poliglactin)
  Interventions: Procedure: Synthetic sling surgery
- Ultrapromesh®(Ethicon,USA) (Active Comparator): Ultrapromesh®(semiabsorbable monofilament mesh;non-absorbable Polypropylene+absorbable polyglecaprone).
  Interventions: Procedure: Synthetic sling surgery
- Prolene light mesh®(Johnson&Johnson,USA) (Active Comparator): Prolene light mesh®(cpp-Condensed monofilament non absorbable polypropylene mesh)
  Interventions: Procedure: Synthetic sling surgery

INTERVENTIONS:
Procedure: Synthetic sling surgery — An incision of inverted A shape was inflicted on the anterior vaginal wall(AVW)of the vagina.The upper part of A shaped incision was formed into an island belonging to the vaginal wall.This patch was 3×4cm in most of the patients.Proximal AVWwas dissected as a flap.Synthetics mesh materials were first sutured onto the upper part of the A on the vaginal island with absorbable vicrly sutures.Then,with 2polypropilen sutures,these meshes were fixed on both the right and left sides of this island in a helical manner to form a suspension and using curved Kishner needles,the prolene sutures were transferred to suprapubic area.These sutures were ligated on the rectus fascia in a crosswise manner.The mobile lower wing was advanced onto the island and was sutured onto the vaginal skin with intermittent sutures using 3-0 monocryl sutures.After cystoscopy,the prolene sutures were ligated crosswise in the suprapubic region.Special attention was paid notto create much tension on the mesh material.

SUMMARY:
The purpose of this study is to determine the clinical results contributions to surgical success,and complications of mixed type of mesh materials as well as prolen mesh materials in sling surgery in a 3 year follow-up the first time in literature.

DETAILED DESCRIPTION:
Broad based double forced sling operations were performed in 144 patients by using 3 different types of mesh materials between 2004 and 2007. Group I consisted of 48 patients in whom Vypromesh® (Ethicon,USA) was used; Group II consisted of 48 patients in whom Ultrapromesh®( Ethicon,USA) and Group III consisted of 48 patients in whom Prolene light mesh® (Johnson&Johnson,USA) was used. The data of the patients and the success of the operation were evaluated based on 24hr pad test, ICIQ-SF scoring, and Korman questionnaire analysis.

Main outcome measures:The Ultrapromesh® synthetic sling procedures have lower complications incidence and higher success rates than the other synthetic slings in 3-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Stress urinary incontinence
* Mix urinary incontinence
* Previous failed anti-incontinence surgery
* Previous gynecologic surgery

Exclusion Criteria:

* Urodynamical detrusor overactivity or impaired bladder activity
* Prolaps of pelvic organ
* Urge incontinence
* Neurogenic bladder
* Bladder outlet obstruction
* Urinary fistula, Pregnancy
* Active urinary or vaginal enfection
* Contraindication to anesthesia
* > 100ml PVR urine volume

Ages: 31 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2004-07; Primary Completion 2007-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
continence rates at three years after surgery | three years after surgery
  Ultrapromesh® with its superior biomechanical characteristics and with its high success rates,low vaginal and urethral extrusion and denovo urgency rates determined in clinical studies,can be reliably and effectively used in sling surgery.

SECONDARY OUTCOMES:
urethral erosion at three years after surgery | three years after surgery
vaginal erosion at three years after surgery | three years after surgery
Denovo urgency at three years after surgery | three years after surgery
urine retantion at three years after surgery | three years after surgery
sutur granuloma at three years after surgery | three years after surgery

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839